CLINICAL TRIAL: NCT02715245
Title: A Home-based Rehabilitation Program in Multiple Chronic Diseases: the RITH Trial
Brief Title: Multiple Chronic Diseases: the RITH Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Almeria (Other)
Collaborators: Torrecárdenas Hospital (Unknown); Almería Health District (Unknown)
Responsible Party: Principal Investigator, Remedios López Liria, PhD., Universidad de Almeria
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CEIC-AL 39/2012
Record Dates: First submitted 2016-01-18; First posted 2016-03-22 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Multiple Chronic Diseases
Keywords: home rehabilitation; Primary Health Care; Physiotherapy; chronic disease
MeSH Terms: conditions — Multiple Chronic Conditions; Chronic Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental Group (Experimental): Patients with multiple chronic disease referred to Mobile Rehabilitation and Physical therapy team (MRPTT) and Nurse-led case Management in the province of Almeria that comply the inclusion criteria; as well as their caregivers.
  Interventions: Procedure: Home-based rehabilitation
- Control Group (No Intervention): Patients with multiple chronic disease and their caregivers belonging to health centers or areas where there is no figure MRPTT or Nurse-led case Management to reach this population

INTERVENTIONS:
Procedure: Home-based rehabilitation — Procedure/Surgery: Home-based rehabilitation In the patient's home, the primarily applied treatment has been physical therapy, seeking to achieve the highest possible functionality and gait training. In more than 25% of cases, health education is conducted for families and caregivers. Thus, consistent with the patient's condition and their tolerance to activity and to exercise their self-care independently, rehabilitation interventions are activated that prevent sequelae derived from functional limitations.
  Arms: Experimental Group

SUMMARY:
In this research, investigators pretent to evaluate the effectiveness of clinical, functional, psychological and social impact of an intervention model based on shared care between the Mobile Rehabilitation and Physical therapy team (MRPTT) and nurse case managers of Primary Care in a sample of patients with multiple chronic diseases (comorbidities) and their caregivers. A non-randomised controlled trial.

DETAILED DESCRIPTION:
The Experimental group consisted of patients with multiple chronic diseases referred to services in the province of Almería that comply the inclusion criteria and their caregivers. Outcome measures: sex, age, location, primary caregiver, disabling process, number and type of categories including by multiple pathologies, personal history, assessment (physical and functional), Barthel Index, Lawton and Brody index, risk of falls, Scale Pfeiffer, social support, caregiver burden, hospital readmissions and length, technical aids. Quality of Life (SF-12) and degree of user satisfaction. Regarding the intervention: date of application, date of assessment, objectives, treatment / intervention techniques, number of sessions, staff time spent.

Control Group: Patients with multiple diseases and their caregivers, belonging to health centers or areas where there is no figure nurse case manager or MRPTT. Registration information will consist of the same assessments, questionnaires and scales that are comparable to the experimental and control groups for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with multiple chronic diseases that are referred to the nurse case managers and home rehabilitation.
* Detected in Hospital or Primary Care.
* To provide informed consent to participate in research.

Exclusion Criteria:

* clinical situation of agony;
* No acceptance of treatment by the patient or family
* Refuse to participate in the study
* Lack of cooperation of the patient or caregiver.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2015-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Activities of daily living (ADLs) | The Barthel Index is assessing a change between initial assessment, at 2, 6 and 12 months
  The Barthel Index to measure functional, activities of daily living (ADLs) (Mahoney and Barthel, 1965).

SECONDARY OUTCOMES:
Risk of falls | Changes between initial assessment, at 2, 6 and 12 months
  The risk of falls (Jonson Down questionnaire)

OTHER OUTCOMES:
Cognitive state | Changes between initial assessment, at 2, 6 and 12 months
  The cognitive state with Pfeiffer Scale (Pfeiffer, 1975)
The Social Support State | Changes between initial assessment, at 2, 6 and 12 months
  The Social Support State ( assessed with the Gijon abbreviated questionnaire)
Hospital readmissions | Hospital readmissions assessment at 12 months
  number of hospital readmissions

CONTACTS AND LOCATIONS:
Locations (1):
- Torrecárdenas Hospital Complex (Almería) and Almería Health District, Almería, Almería, Spain

IPD SHARING:
Plan to Share IPD: No
According to current legislation ( RD 1090/2015 , Decree 439/210 ) and Law 14/2007 on Biomedical and Health Sciences Research, which regulates the process of clinical trials / observational studies, is the responsibility of the investigator to report regularly to the Committee on Ethics in Research Almeria ( Almería CEI ) the progress of the clinical trial / observational study.

REFERENCES:
- [Derived] Vega-Ramirez FA, Lopez-Liria R, Granados-Gamez G, Aguilar-Parra JM, Padilla-Gongora D. Analysis of home-based rehabilitation in patients with motor impairment in primary care: a prospective observational study. BMC Geriatr. 2017 Jul 14;17(1):145. doi: 10.1186/s12877-017-0526-0. PMID 28705187